CLINICAL TRIAL: NCT00194675
Title: Testosterone Replacement and Dutasteride Effectiveness (TRADE)
Brief Title: TRADE-Testosterone Replacement and Dutasteride Effectiveness
Acronym: TRADE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: GlaxoSmithKline (Industry); Seattle Institute for Biomedical and Clinical Research (Other); VA Office of Research and Development (U.S. Federal Agency); Solvay Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Alvin M. Matsumoto, MD, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01166; 01166, 4-2280-V (Other: VA Puget Sound Health Care System Human Subject Division)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Hypogonadism; Benign Prostatic Hyperplasia
Keywords: androgen deficiency; testosterone; Benign Prostatic Hyperplasia; hypogonadism; prostate; BPH
MeSH Terms: conditions — Hypogonadism; Prostatic Hyperplasia | interventions — Dutasteride; Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone gel + oral placebo (Active Comparator): Testosterone 1% gel 7.5 topical daily + placebo dutasteride orally daily
  Interventions: Drug: Testosterone gel; Drug: Placebo dutasteride
- Testosterone gel + oral dutasteride (Active Comparator): Testosterone 1% gel 7.5 topical daily + dutasteride 0.5 mg orally daily
  Interventions: Drug: Dutasteride; Drug: Testosterone gel

INTERVENTIONS:
Drug: Dutasteride — Dutasteride 0.5 mg orally daily
  Other Names: AndroGel
  Arms: Testosterone gel + oral dutasteride
Drug: Testosterone gel — Testosterone gel 7.5 g daily topical
  Other Names: Testim
Drug: Placebo dutasteride — placebo dutasteride orally daily
  Arms: Testosterone gel + oral placebo

SUMMARY:
The purpose of this research study is to determine whether the combination of the male hormone testosterone [T] in gel form and the oral drug dutasteride [D], used to shrink large prostate glands can safely reduce the size of the prostate gland and symptoms of prostate enlargement (called benign prostatic hyperplasia [BPH]) compared to T treatment alone in men with low testosterone (called hypogonadism).

DETAILED DESCRIPTION:
The primary aim of this study is to determine whether correction of hypogonadism using a combination of testosterone and dutasteride spares subjects from increases in prostate size and symptoms of BPH which may be associated with T alone.

We will also determine the effects of changes in serum T and dihydrotestosterone (DHT) on both the hormonal milieu and genetic program within the prostate gland itself. The technology employed will allow us to determine which genes are androgen responsive within each prostate tissue compartment. Together, these data may determine whether the combination of testosterone and dutasteride safely corrects the symptoms of BPH and hypogonadism and minimizes growth stimulus to the prostate at the genetic level. We will also assess the effects of the combination of T and dutasteride on cognitive function.

This is a six-month, double-blind, randomized, placebo-controlled, single-site study of older hypogonadal men with mild to moderate BPH.

Within each treatment group, a sub-group of subjects will undergo additional procedures as part of a Prostate Biopsy sub-study to obtain prostate tissue for hormonal and genetic analyses. Selection of subjects will be based on clinical indication and/or willingness to undergo prostate biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy older men 50 years old or older
* Hypogonadism; low testosterone (total T less than 280 ng/dL on one occasion or an average of equal to or less than 300 ng/dl on two occasions)
* Prostate volume equal to or more than 30 cc by prostate MRI
* Prostate Specific Antigen (PSA) equal to or more than 1.5 ng/mL and equal to or less than 10 ng/mL
* Subjects with a PSA greater than 4.0 ng/ml must have a negative prostate biopsy
* International Prostate Symptom Score (IPSS) greater than or equal to 8 and less than or equal to 20 at screening
* Comply with study procedures for the full 10 months
* No contraindications to MRI

Subjects with symptomatic Benign Prostatic Hyperplasia (BPH) will be recruited from the Urology and General Internal Medicine Clinics at the VA Puget Sound Health Care System and University of Washington Medical Center in Seattle.

Exclusion Criteria:

* A history of prostate or breast cancer
* Invasive therapy for BPH in the past
* History of acute urinary retention in the 3 months prior to screening
* Previous treatment with a 5 alpha-reductase inhibitor (finasteride or dutasteride)
* Medical therapy for BPH within the past month (alpha-blocker, phytotherapy)
* Use of androgenic or antiandrogenic drugs in the past year
* History or evidence of prostate cancer including suspicious DRE or history of high-grade PIN on prostate biopsy.
* Severe systemic illness (renal, liver, cardiac, lung disease, cancer, diabetes)
* Known untreated obstructive sleep apnea
* Hematocrit greater than 52
* Severe skin disease which may interfere with testosterone gel absorption
* Hypersensitivity to any of the drugs used in the study
* History of a bleeding disorder or need for chronic anticoagulation
* Participation in a drug study concurrently or in the last 90 days
* History or current evidence of drug or alcohol abuse within 12 mo.
* Weight more than 300 lbs.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-03; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvin M Matsumoto, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Background] Gruenewald DA, Matsumoto AM. Testosterone supplementation therapy for older men: potential benefits and risks. J Am Geriatr Soc. 2003 Jan;51(1):101-15; discussion 115. doi: 10.1034/j.1601-5215.2002.51018.x. PMID 12534854
- [Background] Yialamas MA, Hayes FJ. Androgens and the ageing male and female. Best Pract Res Clin Endocrinol Metab. 2003 Jun;17(2):223-36. doi: 10.1016/s1521-690x(03)00018-6. PMID 12787549
- [Background] Jin B, Conway AJ, Handelsman DJ. Effects of androgen deficiency and replacement on prostate zonal volumes. Clin Endocrinol (Oxf). 2001 Apr;54(4):437-45. doi: 10.1046/j.1365-2265.2001.01240.x. PMID 11318778
- [Background] Behre HM, Bohmeyer J, Nieschlag E. Prostate volume in testosterone-treated and untreated hypogonadal men in comparison to age-matched normal controls. Clin Endocrinol (Oxf). 1994 Mar;40(3):341-9. doi: 10.1111/j.1365-2265.1994.tb03929.x. PMID 7514512
- [Background] Huggins C, Hodges CV. Studies on prostatic cancer. I. The effect of castration, of estrogen and androgen injection on serum phosphatases in metastatic carcinoma of the prostate. CA Cancer J Clin. 1972 Jul-Aug;22(4):232-40. doi: 10.3322/canjclin.22.4.232. No abstract available. PMID 4625049
- [Background] Bhasin S, Singh AB, Mac RP, Carter B, Lee MI, Cunningham GR. Managing the risks of prostate disease during testosterone replacement therapy in older men: recommendations for a standardized monitoring plan. J Androl. 2003 May-Jun;24(3):299-311. doi: 10.1002/j.1939-4640.2003.tb02676.x. No abstract available. PMID 12721204
- [Background] Morgentaler A, Bruning CO 3rd, DeWolf WC. Occult prostate cancer in men with low serum testosterone levels. JAMA. 1996 Dec 18;276(23):1904-6. PMID 8968017
- [Background] Schatzl G, Madersbacher S, Thurridl T, Waldmuller J, Kramer G, Haitel A, Marberger M. High-grade prostate cancer is associated with low serum testosterone levels. Prostate. 2001 Apr;47(1):52-8. doi: 10.1002/pros.1046. PMID 11304729
- [Background] Thompson IM, Goodman PJ, Tangen CM, Lucia MS, Miller GJ, Ford LG, Lieber MM, Cespedes RD, Atkins JN, Lippman SM, Carlin SM, Ryan A, Szczepanek CM, Crowley JJ, Coltman CA Jr. The influence of finasteride on the development of prostate cancer. N Engl J Med. 2003 Jul 17;349(3):215-24. doi: 10.1056/NEJMoa030660. Epub 2003 Jun 24. PMID 12824459
- [Background] Monti S, Di Silverio F, Iraci R, Martini C, Lanzara S, Falasca P, Poggi M, Stigliano A, Sciarra F, Toscano V. Regional variations of insulin-like growth factor I (IGF-I), IGF-II, and receptor type I in benign prostatic hyperplasia tissue and their correlation with intraprostatic androgens. J Clin Endocrinol Metab. 2001 Apr;86(4):1700-6. doi: 10.1210/jcem.86.4.7413. PMID 11297606
- [Result] Page ST, Hirano L, Gilchriest J, Dighe M, Amory JK, Marck BT, Matsumoto AM. Dutasteride reduces prostate size and prostate specific antigen in older hypogonadal men with benign prostatic hyperplasia undergoing testosterone replacement therapy. J Urol. 2011 Jul;186(1):191-7. doi: 10.1016/j.juro.2011.03.026. Epub 2011 May 14. PMID 21575967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the VA Puget Sound Health Care System, Seattle, WA. 102 men were screened and 53 were randomized.
Pre-assignment Details: 49 were excluded. 4 withdrew consent, 3 lost to follow-up, 42 for inclusion/exclusion criteria: 3 could not tolerate MRI, 3 were previously on testosterone therapy, 21 had prostate volume <30cc, 12 had repeat serum testosterone >280 ng/mL, and 3 had prostate cancer or prostate intraepithelial neoplasia at pre-treatment prostate biopsy.
Groups:
- Testosterone Gel + Oral Placebo: Testosterone 1% topical gel 7.5g daily + placebo dutasteride pill orally daily for 6 months
- Testosterone Gel + Oral Dutasteride: Testosterone 1% topical gel 7.5g daily + dutasteride 0.5 mg orally daily for 6 months
Period: Overall Study
Arm/Group | Testosterone Gel + Oral Placebo | Testosterone Gel + Oral Dutasteride
Started | 27 | 26
Completed | 22 | 24
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — lack of interest | 1 | 1
Not completed — withdrew due to "edgy" feeling | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone Gel + Oral Placebo | Testosterone Gel + Oral Dutasteride | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Customized [Median (Standard Deviation); unit: participants]
  Between 50 and 82 years | 63.5 (8.0) | 63.6 (5.5) | 63.55 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 27 | 26 | 53
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Effects of Testosterone Gel Alone or in Combination With Oral Dutasteride on Prostate Volume in Hypogonadal Men With Benign Prostatic Hyperplasia.
Time Frame: Baseline, Month 6
Population: per protocol
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | Testosterone Gel + Oral Placebo | Testosterone Gel + Oral Dutasteride
Number analyzed (Participants) | 27 | 26
cubic centimeters
  Baseline, Day 0 | 54.2 (38.1) | 44.4 (19.8)
  Month 6 | 58.3 (38.7) | 38.6 (18.4)

2. Secondary Outcome: Serum and Intraprostatic Hormone Levels: Prostate Specific Antigen (PSA)
Time Frame: Baseline, Month 6
Population: per protocol
Measure: Mean (Standard Deviation); unit: ng/ ml
Arm/Group | Testosterone Gel + Oral Placebo | Testosterone Gel + Oral Dutasteride
Number analyzed (Participants) | 27 | 26
ng/ ml
  Baseline PSA | 2.8 (2.9) | 2.1 (1.3)
  Month 6 PSA | 3.1 (2.9) | 1.4 (1.2)

3. Secondary Outcome: The Effects of T Alone or in Combination With Dutasteride on Signs and Symptoms of Benign Prostatic Hyperplasia (BPH) in Hypogonadal Men With Benign Prostatic Hyperplasia. (International Prostate Symptom Score)
Description: International Prostate Symptom Score to assess lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH). Minimum score = 0, maximum score = 35; mildly symptomatic score = 0-7; moderately symptomatic score = 8-19; severely symptomatic score = 20-35; no subscales.
Time Frame: Baseline, Month 3, Month 6
Population: per protocol
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Testosterone Gel + Oral Placebo | Testosterone Gel + Oral Dutasteride
Number analyzed (Participants) | 27 | 26
score
  Baseline IPSS | 13.5 (2.7) | 13.3 (3.1)
  Month 3- IPSS | 11.6 (5.0) | 10.2 (5.4)
  Month 6 IPSS | 11.1 (5.2) | 10.3 (6.6)

4. Secondary Outcome: Signs and Symptoms of Benign Prostatic Hyperplasia (BPH) in Hypogonadal Men (Uroflow)
Time Frame: Baseline, 3-months, 6-months
Population: per protocol
Measure: Mean (Standard Deviation); unit: cc/sec
Groups:
- Testosterone Gel + Oral Placebo: Testosterone 1% gel 7.5 daily + oral placebo dutasteride daily
- Testosterone Gel + Oral Dutasteride: Testosterone 1% gel 7.5 daily + dutasteride 0.5 mg po daily
Arm/Group | Testosterone Gel + Oral Placebo | Testosterone Gel + Oral Dutasteride
Number analyzed (Participants) | 27 | 26
cc/sec
  Baseline Uroflow, Baseline | 13.8 (3.0) | 13.4 (3.5)
  Uroflow after 3 months of treatment | 12.7 (3.4) | 13.2 (5.8)
  Uroflow after 6 months of treatment | 13.8 (5.1) | 14.6 (6.7)

5. Secondary Outcome: Signs and Symptoms Benign Prostatic Hyperplasia (BPH): Post-voiding Residual (PVR) Urinary Volume
Time Frame: Baseline, 3-months, 6-months
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Testosterone Gel + Oral Placebo | Testosterone Gel + Oral Dutasteride
Number analyzed (Participants) | 27 | 26
cc
  Baseline Post Residual Volume (PVR) | 43 (44) | 48 (55)
  3 month Post Residual Volume | 36 (36) | 41 (42)
  6 month Post Residual Volume | 39 (45) | 32 (36)

6. Secondary Outcome: Serum Hormone Levels: Total Testosterone, Free Testosterone, and Dihydrotestosterone(DHT), Dehydroepiandrosterone(DHEA), and Androstenedione.
Time Frame: Baseline, 3-months, 6-months
Population: per protocol
Measure: Mean (Standard Deviation); unit: ng/ dL
Arm/Group | Testosterone Gel + Oral Placebo | Testosterone Gel + Oral Dutasteride
Number analyzed (Participants) | 27 | 26
ng/ dL
  Total testosterone, baseline | 206 (109) | 213 (68)
  Total testosterone, month 3 | 494 (331) | 525 (268)
  Total testosterone, month 6 | 481 (329) | 534 (360)
  Free testosterone, baseline | 4.2 (2.0) | 4.5 (1.8)
  Free testosterone, month 3 | 11.3 (6.8) | 12.0 (6.1)
  Free testosterone, month 6 | 11.4 (11.1) | 12.3 (9.6)
  Dihydrotestosterone (DHT), baseline | 47 (94) | 28 (15)
  Dihydrotestosterone (DHT), month 3 | 145 (120) | 16 (11)
  Dihydrotestosterone (DHT), month 6 | 134 (87) | 12 (7)
  Dehydroepiandrosterone (DHEA), baseline | 72 (42) | 99 (68)
  Dehydroepiandrosterone (DHEA), month 3 | 98 (92) | 109 (93)
  Dehydroepiandrosterone (DHEA), month 6 | 97 (86) | 111 (90)
  Androstenedione, baseline | 45 (21) | 47 (28)
  Androstenedione, month 3 | 99 (72) | 140 (60)
  Androstenedione, month 6 | 100 (57) | 123 (61)

ADVERSE EVENTS:
Time Frame: 4 years. The study was conducted from March 2005 - March 2009.
Arm/Group | Testosterone Gel + Oral Placebo | Testosterone Gel + Oral Dutasteride
Serious Adverse Events (participants affected / at risk) | 2/27 | 0/26
Other Adverse Events (participants affected / at risk) | 7/27 | 4/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Gel + Oral Placebo (N=27) | Testosterone Gel + Oral Dutasteride (N=26)
death from myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — Subject had history of cardiovascular disease prior to randomization and normal hematocrit. Subject died during month 6.
non-ST segment myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — Subject had history of cardiovascular disease prior to randomization and normal hematocrit. Adverse event occurred during month 4.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Gel + Oral Placebo (N=27) | Testosterone Gel + Oral Dutasteride (N=26)
mild breast tenderness (Reproductive system and breast disorders) | 2 (2) | 2 (2)
ezcema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
exacerbation of pre-existing colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
increase in prostate specific antigen (PSA) (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Elevated hematocrit (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — transient rash at gel application site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No